CLINICAL TRIAL: NCT04258436
Title: Serratus Anterior Plane Block for Management of Post Thoracotomy Pain and Facilitation of Early Recovery After Pediatric Cardiac Surgery
Brief Title: Serratus Anterior Plane Block for Management of Post Thoracotomy Pain
Acronym: SAPB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: I believe 1 patient was enrolled. The original PI left the institution and the study was not continued after her departure.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Rania K. Abbasi, Associate Professor of Clinical Anesthesia, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1905162549
Record Dates: First submitted 2019-08-30; First posted 2020-02-06 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Opioid Use; Post-thoracotomy Pain Syndrome; Local Anaesthetic Agent Overdose; Local Anesthetic Complication; Pain, Postoperative
Keywords: Post thoractomy pain; Fascial plane blocks; Early recovery after thoractomy; Serratus anterior fascial block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Pediatric Cardiovascular ICU personnel will be blinded to the randomization assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1-Block Arm (Active Comparator): Group1 will receive an ultra-sound guided serratus anterior block after induction of general anesthesia
  Interventions: Procedure: Serratus anterior block
- Group 2-No Block Arm (No Intervention): Group 2 will not receive a serratus block after induction of general anesthesia

INTERVENTIONS:
Procedure: Serratus anterior block — Serratus anterior block will be performed using an ultrasound guided transducer to inject 2mg/kg of 0.2% ropivacaine
  Arms: Group 1-Block Arm

SUMMARY:
This is a single-center, randomized, prospective study evaluating the effect of serratus anterior plane block performed after induction of anesthesia, but before the start of surgery on postoperative opioid requirements. The hypothesis of the study is that serratus anterior plane blocks are relatively simple to perform, provide good postoperative analgesia, facilitate early tracheal extubation, and reduce the length of hospital stay after pediatric cardiac surgery through a thoracotomy.

DETAILED DESCRIPTION:
This is a single-center, randomized, prospective study evaluating the effect of serratus anterior plane block performed after induction of anesthesia, but before the start of surgery on postoperative opioid requirements. There is already a postoperative protocol for the management of pain in the pediatric cardiac intensive care unit. This protocol will be maintained so all patients will be receiving clinically accepted and standard postoperative pain management.

Routine preoperative evaluation will be performed to establish eligibility for study inclusion. All patients will receive anesthesia by a pediatric cardiac anesthesiologist according to the clinical protocol established for these patients. The serratus anterior plane block will be performed by a pediatric anesthesiologist on the acute pain service team who routinely perform pain blocks at this institution.

Group 1 will receive an ultra-sound guided serratus anterior block after induction of general anesthesia. Group 2 will not receive a serratus anterior block.

Postoperative pain will be managed by a pediatric cardiac intensivist according to a standard pain protocol.

ELIGIBILITY:
Inclusion Criteria:

* 12 months of age or less
* Infants undergoing cardiac surgery through a thoracotomy incision
* Infants having surgery performed by a Pediatric Cardiac Surgeon at Riley Hospital

Exclusion Criteria:

* Infants requiring sternotomy or emergency surgery
* Allergy to local anesthetics
* Neonates less that 37 weeks gestation
* Infants intubated prior to surgery
* Infection at the site of the Serratus Anterior Plane Block 6. Bleeding diathesis with increased risk of hematoma at the block site 7. Allergy to morphine 8. Active pulmonary infection

Ages: 38 Weeks to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Measurement of Postoperative Narcotic Exposure | From start of anesthesia to 24 hours postoperatively
  Total morphine equivalents in first 24 hours

SECONDARY OUTCOMES:
Duration of Mechanical Ventilation | From date and time of endotracheal intubation to the date and time of endotracheal extubation up to 100 days
  Total Time in hours and minutes of endotracheal intubation from date and time of intubation to the date and time of extubation up to 100 days
Length of Cardiovascular ICU stay | From admission to the Cardiovascular ICU until discharge ready time from the Cardiovascular ICU up to 100 days
  Duration of hospital stay in the Cardiovascular ICU in hours up to 100 days
Postoperative Pain Scores | From arrival to ICU to 24 hours postoperatively
  Pain scores reported at arrival to ICU, and at 1, 2, 4, 6,8,10,12,and 24 hours
Duration of Supplemental oxygen exposure | From date and time arriving in the ICU to date and time of discharge from hospital up to 100 days
  Total time of supplemental oxygen usage from date and time of endotracheal extubation and application of supplemental oxygen to date and time of supplemental oxygen discontinuation up to 100 days
Adverse events | From block placement until 72 hours post operatively
  Complications from the block, anesthesia or the surgery up to 72 hours post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Cossu, MD, Principal Investigator — Indiana University Department of Anesthesia
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No